CLINICAL TRIAL: NCT04873635
Title: Patient's Expectation and Satisfaction of Implant-supported Prostheses After Excision of Pathological Jaw Lesions: A Prospective Follow-up Study
Brief Title: Expectation and Satisfaction of Implant Rehab After Jaw Surgery
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Walter Y.H. Lam, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: Ref.1/8/12d
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Missing Teeth
Keywords: dental implants; oral surgical procedures; dental prosthesis, implant-supported; patient reported outcome measures; patient satisfaction; quality of life
MeSH Terms: conditions — Anodontia; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had excised pathological jaw lesions and will receive implant rehabilitation
  Interventions: Other: Implant support prostheses

INTERVENTIONS:
Other: Implant support prostheses — Implant support prostheses was provided to restore the missing teeth and tissues removed due to pathological jaw lesions

SUMMARY:
Objective: The aim of this prospective study was to investigate the patient-reported outcome measures (PROMs) of implant-supported prostheses (ISP) among patients who had excised pathological jaw lesions.

Material and Methods: Patients who met the inclusion/exclusion criteria in a dental teaching hospital were recruited. Data pertaining to sociodemographic factors, conditions requiring surgery, surgical procedures and related complications, and types of ISP were collected. Patients' expectation and satisfaction to the ISP including oral health, self-perceived appearance, speech, chewing ability, oral comfort and ease of cleaning were assessed using the visual analogue scale (VAS, 0-100) and global transitional scale/judgement (Likert scale). Data were analysed using t-test and chi-square tests at the significance level α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received surgical removal of pathological jaw lesions in Queen Mary Hospital
* Subjects who plan to receive implant-supported prostheses in Prince Philip Dental Hospital

Exclusion Criteria:

* Subjects with debilitating illnesses or complicating medical conditions
* Subjects who under age of 18 or unable to give consent
* Subjects with uncontrolled caries and periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had received surgical removal of pathological jaw lesions in a university teaching hospital, Queen Mary Hospital, and planned to receive implant-supported reconstruction in a dental teaching hospital, Prince Philip Dental Hospital, Hong Kong, China were recruited
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Patient expectation of implant-supported prosthesis | Before receive implant-supported prosthesis (baseline)
  Visual analogue scale 0-100 which 0 is "No expectation" and 100 is "High expectation"
  Assess general satisfaction, appearance, speech, chewing hard/soft/fibrous foods, comfort, cleaning, occlusion, stability and in comparison to natural teeth
Patient satisfaction of implant-supported prosthesis in 3-point Likert transition scale | Before (baseline) and 3 months post-insertion of implant-supported prosthesis
  Assess changes in oral condition, appearance, speech, chewing hard/soft/fibrous foods, oral comfort and cleaning following jaw surgery and oral rehabilitation
  Global transition judgements: Better, No difference, Worse
Patient satisfaction of implant-supported prosthesis in 0-100 visual analogue scale | 3 months post-insertion of implant-supported prosthesis
  Visual analogue scale 0-100 which 0 is totally unsatisfied and 100 is totally satisfied
  Assess oral health, appearance, speech, chewing hard/soft/fibrous foods, comfort, cleaning, occlusion, and the ability to chew and bite
Patient satisfaction of implant-supported prosthesis in 5-point Likert scale | 3 months post-insertion of implant-supported prosthesis
  Assess
  1. Feeling of health of own teeth, lips, jaw and mouth Global transition scales: Very good, Good, Fair, Poor, Very Poor
  2: Extent of oral health affecting overall life Global transition scales: Very much, A lot, Some, Very little, Not at all

CONTACTS AND LOCATIONS:
Overall Officials: Walter Lam, Principal Investigator — Faculty of Dentistry, The University of Hong kong

IPD SHARING:
Plan to Share IPD: No
Data will be share upon request

REFERENCES:
- [Background] Allen PF, O'Sullivan M, Locker D. Determining the minimally important difference for the Oral Health Impact Profile-20. Eur J Oral Sci. 2009 Apr;117(2):129-34. doi: 10.1111/j.1600-0722.2009.00610.x. PMID 19320721
- [Background] Baracat LF, Teixeira AM, dos Santos MB, da Cunha Vde P, Marchini L. Patients' expectations before and evaluation after dental implant therapy. Clin Implant Dent Relat Res. 2011 Jun;13(2):141-5. doi: 10.1111/j.1708-8208.2009.00191.x. PMID 19681923
- [Background] Gurlek A, Miller MJ, Jacob RF, Lively JA, Schusterman MA. Functional results of dental restoration with osseointegrated implants after mandible reconstruction. Plast Reconstr Surg. 1998 Mar;101(3):650-5; discussion 656-9. doi: 10.1097/00006534-199803000-00011. PMID 9500381
- [Background] Heydecke G, Thomason JM, Awad MA, Lund JP, Feine JS. Do mandibular implant overdentures and conventional complete dentures meet the expectations of edentulous patients? Quintessence Int. 2008 Nov;39(10):803-9. PMID 19093056
- [Background] Hundepool AC, Dumans AG, Hofer SO, Fokkens NJ, Rayat SS, van der Meij EH, Schepman KP. Rehabilitation after mandibular reconstruction with fibula free-flap: clinical outcome and quality of life assessment. Int J Oral Maxillofac Surg. 2008 Nov;37(11):1009-13. doi: 10.1016/j.ijom.2008.05.021. Epub 2008 Jul 26. PMID 18657394
- [Background] Iizuka T, Hafliger J, Seto I, Rahal A, Mericske-Stern R, Smolka K. Oral rehabilitation after mandibular reconstruction using an osteocutaneous fibula free flap with endosseous implants. Factors affecting the functional outcome in patients with oral cancer. Clin Oral Implants Res. 2005 Feb;16(1):69-79. doi: 10.1111/j.1600-0501.2004.01076.x. PMID 15642033
- [Background] Jacobsen HC, Wahnschaff F, Trenkle T, Sieg P, Hakim SG. Oral rehabilitation with dental implants and quality of life following mandibular reconstruction with free fibular flap. Clin Oral Investig. 2016 Jan;20(1):187-92. doi: 10.1007/s00784-015-1487-3. Epub 2015 May 12. PMID 25963720
- [Background] Janzen JA, Silvius J, Jacobs S, Slaughter S, Dalziel W, Drummond N. What is a health expectation? Developing a pragmatic conceptual model from psychological theory. Health Expect. 2006 Mar;9(1):37-48. doi: 10.1111/j.1369-7625.2006.00363.x. PMID 16436160
- [Result] Kim HY. Statistical notes for clinical researchers: effect size. Restor Dent Endod. 2015 Nov;40(4):328-31. doi: 10.5395/rde.2015.40.4.328. Epub 2015 Oct 2. No abstract available. PMID 26587420
- [Result] King MT. A point of minimal important difference (MID): a critique of terminology and methods. Expert Rev Pharmacoecon Outcomes Res. 2011 Apr;11(2):171-84. doi: 10.1586/erp.11.9. PMID 21476819
- [Result] Kramer FJ, Dempf R, Bremer B. Efficacy of dental implants placed into fibula-free flaps for orofacial reconstruction. Clin Oral Implants Res. 2005 Feb;16(1):80-8. doi: 10.1111/j.1600-0501.2004.01040.x. PMID 15642034
- [Result] Leung AC, Cheung LK. Dental implants in reconstructed jaws: patients' evaluation of functional and quality-of-life outcomes. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):127-34. PMID 12608678
- [Result] Li X, Zhu K, Liu F, Li H. Assessment of quality of life in giant ameloblastoma adolescent patients who have had mandible defects reconstructed with a free fibula flap. World J Surg Oncol. 2014 Jul 8;12:201. doi: 10.1186/1477-7819-12-201. PMID 25004805
- [Result] Locker D. Measuring oral health: a conceptual framework. Community Dent Health. 1988 Mar;5(1):3-18. No abstract available. PMID 3285972
- [Result] Locker D. Issues in measuring change in self-perceived oral health status. Community Dent Oral Epidemiol. 1998 Feb;26(1):41-7. doi: 10.1111/j.1600-0528.1998.tb01923.x. PMID 9511841
- [Result] Nordenram G, Davidson T, Gynther G, Helgesson G, Hultin M, Jemt T, Lekholm U, Nilner K, Norlund A, Rohlin M, Sunnegardh-Gronberg K, Tranaeus S. Qualitative studies of patients' perceptions of loss of teeth, the edentulous state and prosthetic rehabilitation: a systematic review with meta-synthesis. Acta Odontol Scand. 2013 May-Jul;71(3-4):937-51. doi: 10.3109/00016357.2012.734421. Epub 2012 Oct 29. PMID 23101439
- [Result] Ooi A, Feng J, Tan HK, Ong YS. Primary treatment of mandibular ameloblastoma with segmental resection and free fibula reconstruction: achieving satisfactory outcomes with low implant-prosthetic rehabilitation uptake. J Plast Reconstr Aesthet Surg. 2014 Apr;67(4):498-505. doi: 10.1016/j.bjps.2014.01.005. Epub 2014 Jan 15. PMID 24508227
- [Result] Pappalardo M, Tsao CK, Tsang ML, Zheng J, Chang YM, Tsai CY. Long-term outcome of patients with or without osseointegrated implants after resection of mandibular ameloblastoma and reconstruction with vascularized bone graft: Functional assessment and quality of life. J Plast Reconstr Aesthet Surg. 2018 Jul;71(7):1076-1085. doi: 10.1016/j.bjps.2018.03.008. Epub 2018 Mar 28. PMID 29656899
- [Result] Parbo N, Murra NT, Andersen K, Buhl J, Kiil B, Norholt SE. Outcome of partial mandibular reconstruction with fibula grafts and implant-supported prostheses. Int J Oral Maxillofac Surg. 2013 Nov;42(11):1403-8. doi: 10.1016/j.ijom.2013.05.007. Epub 2013 Jun 15. PMID 23773236
- [Result] Pjetursson BE, Karoussis I, Burgin W, Bragger U, Lang NP. Patients' satisfaction following implant therapy. A 10-year prospective cohort study. Clin Oral Implants Res. 2005 Apr;16(2):185-93. doi: 10.1111/j.1600-0501.2004.01094.x. PMID 15777328
- [Result] Pommer B, Zechner W, Watzak G, Ulm C, Watzek G, Tepper G. Progress and trends in patients' mindset on dental implants. I: level of information, sources of information and need for patient information. Clin Oral Implants Res. 2011 Feb;22(2):223-9. doi: 10.1111/j.1600-0501.2010.02035.x. Epub 2010 Nov 19. PMID 21087319
- [Result] Rogers SN, Devine J, Lowe D, Shokar P, Brown JS, Vaugman ED. Longitudinal health-related quality of life after mandibular resection for oral cancer: a comparison between rim and segment. Head Neck. 2004 Jan;26(1):54-62. doi: 10.1002/hed.10351. PMID 14724907
- [Result] Chang YM, Wallace CG, Hsu YM, Shen YF, Tsai CY, Wei FC. Outcome of osseointegrated dental implants in double-barrel and vertically distracted fibula osteoseptocutaneous free flaps for segmental mandibular defect reconstruction. Plast Reconstr Surg. 2014 Nov;134(5):1033-1043. doi: 10.1097/PRS.0000000000000623. PMID 25054246
- [Result] Rustemeyer J, Bremerich A. Patients' knowledge and expectations regarding dental implants: assessment by questionnaire. Int J Oral Maxillofac Surg. 2007 Sep;36(9):814-7. doi: 10.1016/j.ijom.2007.05.003. Epub 2007 Jul 2. PMID 17604967
- [Result] Shpitzer T, Neligan PC, Gullane PJ, Freeman JE, Boyd BJ, Rotstein LE, Brown DH, Irish JC, Gur E. Oromandibular reconstruction with the fibular free flap. Analysis of 50 consecutive flaps. Arch Otolaryngol Head Neck Surg. 1997 Sep;123(9):939-44. doi: 10.1001/archotol.1997.01900090051007. PMID 9305243
- [Result] Tepper G, Haas R, Mailath G, Teller C, Zechner W, Watzak G, Watzek G. Representative marketing-oriented study on implants in the Austrian population. I. Level of information, sources of information and need for patient information. Clin Oral Implants Res. 2003 Oct;14(5):621-33. doi: 10.1034/j.1600-0501.2003.00916.x. PMID 12969367
- [Result] Vayvada H, Mola F, Menderes A, Yilmaz M. Surgical management of ameloblastoma in the mandible: Segmental mandibulectomy and immediate reconstruction with free fibula or deep circumflex iliac artery flap (evaluation of the long-term esthetic and functional results). J Oral Maxillofac Surg. 2006 Oct;64(10):1532-9. doi: 10.1016/j.joms.2005.11.065. PMID 16982313
- [Result] Vermylen K, Collaert B, Linden U, Bjorn AL, De Bruyn H. Patient satisfaction and quality of single-tooth restorations. Clin Oral Implants Res. 2003 Feb;14(1):119-24. doi: 10.1034/j.1600-0501.2003.140116.x. PMID 12562374
- [Result] Voutilainen A, Pitkaaho T, Kvist T, Vehvilainen-Julkunen K. How to ask about patient satisfaction? The visual analogue scale is less vulnerable to confounding factors and ceiling effect than a symmetric Likert scale. J Adv Nurs. 2016 Apr;72(4):946-57. doi: 10.1111/jan.12875. Epub 2015 Dec 22. PMID 26689434
- [Result] Yao J, Tang H, Gao XL, McGrath C, Mattheos N. Patients' expectations to dental implant: a systematic review of the literature. Health Qual Life Outcomes. 2014 Oct 29;12:153. doi: 10.1186/s12955-014-0153-9. PMID 25358599
- [Result] Zhu J, Yang Y, Li W. Assessment of quality of life and sociocultural aspects in patients with ameloblastoma after immediate mandibular reconstruction with a fibular free flap. Br J Oral Maxillofac Surg. 2014 Feb;52(2):163-7. doi: 10.1016/j.bjoms.2013.10.012. Epub 2013 Nov 23. PMID 24280117